CLINICAL TRIAL: NCT03023956
Title: Outcome of Proximal Humerus Fractures :Anatomic Neck Fractures vs Surgical Neck Fractures
Status: Completed | Type: Observational
Sponsor: Xiaoxiao Zhou (Other)
Responsible Party: Sponsor-Investigator, Xiaoxiao Zhou, Professor, Zhoupu Hospital, Pudong New Area, Shanghai, China
Organization: Zhoupu Hospital, Pudong New Area, Shanghai, China (Other)
Other Study IDs: ZhouXuANFSNF
Record Dates: First submitted 2017-01-12; First posted 2017-01-18 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Humeral Fracture, Proximal; Internal Fixation; Complications, Mechanical, Bones of Limb
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- ANF: anatomic neck fractures of proximal humerus
  Interventions: Procedure: Locking plates were used for proximal humeral fractures.
- SNF: surgical neck fractures of proximal humerus
  Interventions: Procedure: Locking plates were used for proximal humeral fractures.

INTERVENTIONS:
Procedure: Locking plates were used for proximal humeral fractures.

SUMMARY:
From April ,2014 to April 2015,31 patients with fractures of the proximal humerus were treated in our hospital. According to anatomic neck fractures (ANF) and surgical neck fractures (SNF), we divided the patients into two groups. All the patients were followed at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

-From May ,2013 to April 2015, patients with fractures of the proximal humerus who were treated with locking plate.

Exclusion Criteria:

* Patients had pathologic fractures,
* Patients had previous surgery on the affected shoulder,
* Patients were treated with shoulder arthroplasty.
* Patients were treated with intramedullary nail.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From May ,2013 to April 2015, patients with fractures of the proximal humerus who were treated with locking plate.
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2016-07; Primary Completion 2016-12 (Actual); Study Completion 2017-01-03 (Actual)

PRIMARY OUTCOMES:
change of head-shaft angle at 12months from 6months in two groups | 12months

SECONDARY OUTCOMES:
change of Offset at 12months from 6months in two groups | 12 months
Constant-Murly scores at 3 months, 12 months and last follow-up | 3 months,12 months,last follow-up (last follow-up means recent evaluation before database lock, it is more than 12months )
change of the distance between the screw tip and the subchondral surface(TSD) at 12months from 6months in two groups | 12 months